CLINICAL TRIAL: NCT01757470
Title: Effectiveness of Risk Minimisation Interventions for Vandetanib in Canada
Brief Title: Vandetanib Risk Minimisation Effectiveness
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: D4200L00059
Record Dates: First submitted 2012-12-18; First posted 2012-12-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Medullary Thyroid Cancer
Keywords: effectiveness of risk mitigation,; knowledge and understanding survey,; drug utilisation study,; post marketing commitments
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Caprelsa Patient: All patients treated with Caprelsa in Canada and participating in the restricted distribution programme.
- Caprelsa Prescriber: All physicians having prescribed at least one dose of Caprelsa and registered as a certified prescriber of Caprelsa in Canada.

SUMMARY:
Effectiveness of risk minimisation interventions for vandetanib in Canada

DETAILED DESCRIPTION:
As part of the new drug approval process in Canada, AstraZeneca has committed to Health Canada to conduct a Drug Utilization Study among patients recently treated with CAPRELSA (vandetanib) and a Knowledge and Understanding Survey among the prescribing physicians to determine whether the product monograph, communication plan, and educational material developed by AstraZeneca Canada for vandetanib are adequate to provide knowledge about the potential risks associated with this product, and if other medications taken concomitantly with vandetanib are managed adequately.

ELIGIBILITY:
Inclusion Criteria:

- N/A (all patients taking Caprelsa and all prescribers will be contacted for participation).

Exclusion Criteria: - N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Convenience sample for patients and physicians
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Knowledge and Understanding Survey: Knowledge of the key safety issues pertaining to vandetanib | 2 months
  QT prolongation/TdP Torsades, diarrhea, rash and other skin reactions- adequate or inadequate for each safety issue (defined by correct response).
Drug Utilisation Study: Use of vandetanib - duration of treatment at baseline | At baseline
  Discontinuation, interruption, continuous
Drug Utilisation Study: Use of vandetanib - duration of treatment at 3 months | At 3 months
  Discontinuation, interruption, continuous
Drug Utilisation Study: Use of vandetanib - duration of treatment at 6 months | At 6 months
  Discontinuation, interruption, continuous
Drug Utilisation Study: Use of vandetanib - duration of treatment at 12 months | At 12 months
  Discontinuation, interruption, continuous
Drug Utilisation Study: Use of vandetanib - dosage at baseline | At baseline
Drug Utilisation Study: Use of vandetanib - dosage at 3 months | At 3 months
Drug Utilisation Study: Use of vandetanib - dosage at 6 months | At 6 months
Drug Utilisation Study: Use of vandetanib - dosage at 12 months | At 12 months
Drug Utilisation Study: Concomitant use of QT-prolonging drugs at baseline | At baseline
  Dichotomous variable - yes/no + total number of concomitant QT-prolonging drugs
Drug Utilisation Study: Concomitant use of QT-prolonging drugs at 3 months | At 3 months
  Dichotomous variable - yes/no + total number of concomitant QT-prolonging drugs
Drug Utilisation Study: Concomitant use of QT-prolonging drugs at 6 months | At 6 months
  Dichotomous variable - yes/no + total number of concomitant QT-prolonging drugs
Drug Utilisation Study: Concomitant use of QT-prolonging drugs at 12 months | At 12 months
  Dichotomous variable - yes/no + total number of concomitant QT-prolonging drugs

SECONDARY OUTCOMES:
Knowledge and Understanding Survey: Practice characteristics | 2 months
  Main geographical location, average days devoted to patient care, total number of medullary thyroid cancer patients followed up to date.
Knowledge and Understanding Survey: Previous exposure to vandetanib safety concerns other than product monograph or mandatory online training | 2 months
  Participation in a trial on vandetanib, giving CME conferences, member of a data safety monitoring board.
Knowledge and Understanding Survey: Sources of information on key safety messages for vandetanib | 2 months
  Product monograph, online training, Dear Healthcare Professional letter sent by AstraZeneca, company's sales forces, continuing medical education, conferences.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Research Site, Montreal, Quebec, Canada